CLINICAL TRIAL: NCT00773357
Title: Modeling Stress-precipitated Smoking Behavior for Medication Development
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Office of Research on Women's Health (ORWH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sherry McKee, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0808004163; RL1DA024857 (NIH); P50DA033945 (NIH); P01AA027473 (NIH); U54AA027989 (NIH)
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Results first posted 2022-08-01 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Smoking
Keywords: smoking lapse behavior; guanfacine
MeSH Terms: conditions — Smoking | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guanfacine (Experimental): guanfacine 3mg/day
  Interventions: Drug: guanfacine
- Placebo (Placebo Comparator): placebo control
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: guanfacine — 3 mg/day, with 3-week lead-in medication period. The starting dose is 0.5 mg/day for days 1-3, followed by 1.5mg/day for days 4-7, followed by 2 mg/day for days 8-12, followed by 2.5 mg/day for days 13-15, followed by 3 mg/day from day 16 to remainder of study. 5-day taper at end of study.
  Other Names: Tenex
  Arms: Guanfacine
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine whether guanfacine will attenuate the ability of stress to precipitate smoking lapse behavior in treatment seeking and non-treatment seeking daily smokers.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-60
* able to read and write in English
* smokers

Exclusion Criteria:

* any significant current medical conditions that would contraindicate smoking
* current Diagnostic and Statistical Manual IV (DSM-IV) abuse or dependence of other substances, other than nicotine (or caffeine) dependence
* positive test result at intake appointments on urine drug screens conducted for opiates, cocaine, or benzodiazepines
* women who are pregnant or nursing
* suicidal, homicidal or evidence of severe mental illness
* participants prescribed any psychotropic drug in the 30 days prior to study enrollment
* blood donation within the past 6 weeks
* participants who have engaged in a quit attempt in the past 3 months
* specific exclusions for administration of guanfacine not already specified include: Hypotensive individuals with sitting blood pressure below 90/50 mmHG; EKG evidence at baseline screening of any clinically significant conduction abnormalities, including a Bazett's corrected QT interval (QTc) >450 msec for men and QTc>470 msec for women; known intolerance for guanfacine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-10; Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation, Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Guanfacine | Placebo
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guanfacine | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.36 (10.05) | 36.92 (11.73) | 36.14 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 27 | 28 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 18 | 31
  White | 32 | 28 | 60
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 15.44 (7.58) | 15.12 (8.11) | 15.28 (7.845)

OUTCOME MEASURES:

1. Primary Outcome: Latency to Initiate Ad-lib Smoking Session
Description: latency to initiate smoking (in minutes) during a 50-minute period.
Time Frame: 50 minutes
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Guanfacine | Placebo
Number analyzed (Participants) | 50 | 50
minutes | 31.55 (5.30) | 30.31 (5.44)

ADVERSE EVENTS:
Time Frame: Titration period of 21 days
Arm/Group | Guanfacine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 35/50 | 12/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guanfacine (N=50) | Placebo (N=50)
dry mouth (General disorders) | 35 | 12
Drowsiness (General disorders) | 19 | 9
Dizziness (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 15 | 10
Impotence (Reproductive system and breast disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 10 | 6
Fatigue (General disorders) | 18 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/57/NCT00773357/Prot_SAP_000.pdf